CLINICAL TRIAL: NCT06728488
Title: Comparison of the Analgesic Efficacy and Duration of Analgesic Effect of PENG Block Application With PENG Block and Pulse Radiofrequency Ablation in Chronic Hip Pain
Brief Title: Comparison of the Analgesic Efficacy and Duration of Analgesic Effect of Pericapsular Nerve Group Block Block Application With PENG Block and Pulse Radiofrequency Ablation in Chronic Hip Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Collaborators: Scientific Research Projects Coordination Unit (Ambiguous)
Responsible Party: Principal Investigator, Berkay BALCI, Research Assistant Doctor, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AIBU-MED-BB-01
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Hip Pain Chronic
Keywords: hip pain chronic; Radiofrequency ablation; PENG block; vNRS (Verbal Numerical Rating Scale)

STUDY DESIGN:
Intervention Model Description: Comparison of the analgesic efficacy and duration of analgesic effect of PENG block application with PENG block and pulse radiofrequency ablation in chronic hip pain.
Who Masked: Participant
Masking Description: Both surgical groups will be randomly assigned into groups using simple randomization through the -www.randomize.net- application, and a single-blind design will be implemented.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG block (Experimental): The patients in the PENG block group will provide their consent. Standard monitoring will be applied. The patients will be positioned supine. After antiseptic procedures, 2 ml of 2% lidocaine will be infiltrated into the needle insertion site. The linear ultrasound probe will be placed in the transverse plane over the AIIS. The position of the ultrasound probe will be verified by visualizing the iliopectineal eminence, iliopsoas muscle and tendon, femoral artery, and pectineus muscle. Using a Stimuplex® A 100 mm 20 gauge needle (Braun Melsungen AG, Melsungen, Germany) with the in-plane technique, the needle will be inserted laterally to medially into the space between the psoas tendon and the pubic ramus. Negative aspiration will be performed to ensure no blood is aspirated, and then 20 ml of 0.25% bupivacaine and 8 mg of dexamethasone will be injected to perform the PENG block. After the procedure, the cannula will be removed, and the insertion site will be cleaned and dressed.
  Interventions: Other: PENG Block
- PENG block and pulse radiofrequency ablation (Experimental): After obtaining consent, the patients in the PENG block and pulse radiofrequency ablation group will be brought into the operating room. Standard monitoring will be applied (ECG, SpO2, NIBP). The patients will be positioned supine. After performing the necessary aseptic and antiseptic procedures, 2 ml of 2% lidocaine will be infiltrated into the needle insertion site. The Boston Scientific unified echogenic 10cmx10mmx20G (0.9mm) radiofrequency cannula will be advanced until it makes contact with the superior ramus near the iliopectineal eminence. Pulse radiofrequency ablation will be performed with two cycles of 90 seconds each, and after each cycle, the needle will be moved 2 mm medially. After pulse radiofrequency ablation, 20 ml of 0.25% bupivacaine and 8 mg of dexamethasone will be applied. After the procedure, the cannula will be removed, and the insertion site will be cleaned and dressed.
  Interventions: Other: PENG block and pulse radiofrequency ablation

INTERVENTIONS:
Other: PENG Block — The patients in the PENG block group will provide their consent. Standard monitoring will be applied. The patients will be positioned supine. After antiseptic procedures, 2 ml of 2% lidocaine will be infiltrated into the needle insertion site. The linear ultrasound probe will be placed in the transverse plane over the AIIS. The position of the ultrasound probe will be verified by visualizing the iliopectineal eminence, iliopsoas muscle and tendon, femoral artery, and pectineus muscle. Using a Stimuplex® A 100 mm 20 gauge needle (Braun Melsungen AG, Melsungen, Germany) with the in-plane technique, the needle will be inserted laterally to medially into the space between the psoas tendon and the pubic ramus. Negative aspiration will be performed to ensure no blood is aspirated, and then 20 ml of 0.25% bupivacaine and 8 mg of dexamethasone will be injected to perform the PENG block. After the procedure, the cannula will be removed, and the insertion site will be cleaned and dressed.
  Arms: PENG block
Other: PENG block and pulse radiofrequency ablation — After obtaining consent, the patients in the PENG block and pulse radiofrequency ablation group will be brought into the operating room. Standard monitoring will be applied (ECG, SpO2, NIBP). The patients will be positioned supine. After performing the necessary aseptic and antiseptic procedures, 2 ml of 2% lidocaine will be infiltrated into the needle insertion site. The Boston Scientific unified echogenic 10cmx10mmx20G (0.9mm) radiofrequency cannula will be advanced until it makes contact with the superior ramus near the iliopectineal eminence. Pulse radiofrequency ablation will be performed with two cycles of 90 seconds each, and after each cycle, the needle will be moved 2 mm medially. After pulse radiofrequency ablation, 20 ml of 0.25% bupivacaine and 8 mg of dexamethasone will be applied. After the procedure, the cannula will be removed, and the insertion site will be cleaned and dressed.
  Arms: PENG block and pulse radiofrequency ablation

SUMMARY:
Comparison of the analgesic efficacy and duration of analgesic effect of PENG block application with PENG block and pulse radiofrequency ablation in chronic hip pain.

DETAILED DESCRIPTION:
Patients with chronic hip pain will be divided into two groups, and after providing the necessary information, informed consent forms will be obtained for inclusion in the study from both groups. The 'Verbal Numerical Rating Scale (vNRS)' will be assessed before the procedure. Patients to undergo PENG block and PENG block with pulse radiofrequency ablation will be monitored prior to the procedure. After the procedure, they will be monitored for 3 hours under observation. At the third hour after the procedure, before leaving the operating room, and at the 1st and 3rd months, patients will be contacted by phone, and the 'Verbal Numerical Rating Scale (vNRS)' will be evaluated. This will allow the comparison of the effects of PENG block and PENG block with pulse radiofrequency ablation on pain management in chronic hip pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic hip pain Aged 18-80 ASA I-III patients

Exclusion Criteria:

* Patients with allergies to the medications used, severe cardiac, renal, pulmonary, liver, and endocrine diseases, patients with uncontrolled blood sugar levels (diabetes mellitus), patients who have used anticoagulant medications in the last five days, patients with bleeding or clotting disorders, those with implanted medical devices such as pacemakers and defibrillators, patients with infections at the procedure site, patients with psychiatric disorders or communication difficulties, patients with missing data, and patients who do not wish to undergo regional block are defined as exclusion criteria.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
vNRS Verbal Numerical Rating Scale | 3 months
  Verbal Numerical Rating Scale.At the 3rd hour after the procedure, before the patients leave the operating room, and at the 1st and 3rd months, they will be contacted by phone, and the 'Verbal Numerical Rating Scale (vNRS)' will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, IZMIT, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes